CLINICAL TRIAL: NCT03548831
Title: Comparative Study of Laparoscopic Assisted Vaginal Hysterectomy and Minilap Hysterectomy for Benign Gynaecological Conditions
Brief Title: Comparative Study of LAVH and Minilaparotomy Hysterectomy
Acronym: LAVH
Status: Completed | Type: Observational
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Abhilasha Agarwal, Junior Resident, Manipal University
Other Study IDs: IEC 429/2014
Record Dates: First submitted 2018-04-16; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Hysterectomy; Minimal Invasive Surgery; Benign Gynecologic Neoplasm
Keywords: Minilaparotomy; Hysterectomy; Laparoscopic assisted vaginal hysterectomy; Benign; Gynaecology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MLH: Minilaparotomy Hysterectomy
- LAVH: Laparoscopic Assisted Vaginal Hysterectomy

SUMMARY:
Minilaparotomy hysterectomy (MLH) relies on the simplicity of traditional open technique of abdominal hysterectomy, imparts cosmesis and faster recovery of laparoscopic hysterectomy yet avoids the long learning curve, cost of expensive setup and instrumentation associated with the minimally invasive approaches namely laparoscopy and robotics. In the present study, we tried to ascertain if the results obtained with MLH can be compared to LAVH in terms of its feasibility, intraoperative variables, and complications. The null hypothesis was that both MLH and LAVH are comparable techniques, so where cost and surgeon's experience are the confining issues, patients can be reassured that MLH gives comparable results.

DETAILED DESCRIPTION:
Around 600,000 hysterectomies are performed every year in the United States, making hysterectomy the second most common surgery for women, first being cesarean section. Most of the hysterectomies are done for non cancerous conditions. And the most common indication for the same is symptomatic fibroid uterus.

In spite of being the most common gynaecological surgery the route of hysterectomy has always been an issue of debate since early 19th century. In the beginning it started as vaginal hysterectomy which soon was taken over by laparotomy route. With the advent of laparoscopy as the recent minimally invasive route the choices have further increased. Laparoscopic route has prompted the need for development of other forms of hysterectomy which are minimally invasive and are associated with less perioperative morbidity with better postoperative outcomes. Abdominal route includes both conventional and minilaparotomy; laparoscopic route includes both Laparoscopic Assisted Vaginal Hysterectomy (LAVH) as well as Total Laparoscopic Hysterectomy (TLH). Each method has its own advantages and disadvantages. The vaginal route is preferable because it is associated with less perioperative morbidity and faster recovery. Although laparoscopic route offers minimally invasive alternative to abdominal hysterectomy when vaginal route is contraindicated (In case of huge fibroid uterus or patients with pelvic pathology), it has its own drawbacks. The laparoscopic instruments are costly, there is a long learning curve involved in the training, and the operating time with this route is prolonged.

The EVALUATE study suggested that majority of surgeons(67%) preferred abdominal approach as the route of surgery, especially when dealing with pelvic pathology. Hence, minilaparotomy hysterectomy as an alternative minimally invasive surgery method was started. It relies on traditional open techniques and inexpensive instrumentation, making it significantly faster than laparoscopy and easy to perform. Hoffman et al found minilaparotomy hysterectomy procedure effective and safe in non-obese women in whom vaginal approach was contraindicated. Fanfani et al did a retrospective analysis on 252 patients who underwent minilaparotomy hysterectomy and found it to be a feasible route of surgery in benign gynaecological conditions with operative time similar or shorter as compared to vaginal, laparotomy and laparoscopy surgery. Few surgeons have modified the incision depending on the their experience which led to development of Pelosi method of Minilaparotomy Hysterectomy in 2003.

The final choice of the route and method depends on multiple factors which include indication of surgery, size of fibroid, equipments available in the surgical set up, surgeons' expertise, patient's financial background.

All patients followed the same standard pre-operative protocol. All surgeries were performed under general anesthesia with endotracheal intubation. Demographic details that included age, parity, body mass index (BMI), baseline investigations, diagnosis, and co-morbidities, were collated a day prior to the day of surgery. On admission, patients were informed in detail about the operation modalities and the associated complications. Patients along with their relatives were counselled about the advantages and disadvantages of both the surgical methods and the final decision was made on a joint consensus between the surgeon and the patient, following which an informed written consent was obtained.

The aim of the study was to compare the feasibility of two minimally invasive surgical procedures in low resource settings (such as India) - Laparoscopic assisted vaginal hysterectomy (LAVH) and Minilaparotomy hysterectomy (transverse suprapubic incision <7cm).

ELIGIBILITY:
Inclusion Criteria:

* Non descent uterus with benign gynaecological conditions

Exclusion Criteria:

* Uterine size > 20 weeks
* Minilaparotomy was contraindicated in patients where severe adhesions might exist eg -

  * Endometriosis
  * Previous pelvic inflammatory disease
* Patients with one or more contraindications for LAVH were excluded -

  * Cardiac or respiratory morbidity contraindicating laparoscopy
  * Frozen pelvis
  * Cervix flushed with vagina

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Benign gynaecological conditions
Study Population: Women who are admitted in the Department of OBG, Kasturba Hospital, Manipal for hysterectomy for benign gynaecological disorders with non descent uterus.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Duration of surgery | Intra operatively
  All surgeries were performed by two gynecologists with an almost equal level of surgical competence.
Blood loss | Intra operatively
  Total amount of blood loss was calculated during both the methods. It was calculated by adding up the mop count (one fully soaked mop ~ 50 ml of blood loss) and the amount of fluid in the suction pump minus the saline used for irrigation.
Postoperative pain | Starting from immediate post-operative period till 72 hours.
  There are various methods to score pain. In our study, we used visual analogue scale for the scoring. The pain was scored every 6th hourly for the first 24hrs and thereafter 24th hourly till 72 hrs.
  The Visual Analogue Scale (VAS) (Figure 14) is a scoring scale on which the patient rates his/her pain on a scale of 0 to 10, 0 representing no pain and 10 representing excruciating or intolerable pain. The scoring is subjective and gives the patient freedom to choose the intensity of the pain as per their perception.

SECONDARY OUTCOMES:
Weight of uterus | Intra operatively
  In grams unit
Intra-operative complications | Intra-operatively
  Visceral injury such as bladder/ ureter / bowel injury
Conversion rate | Intraoperatively
  Conversion to conventional laparotomy
Post operative complications | Upto 1 month
  Secondary haemorrhage, Urinary Tract Infection, Urinary retention, Wound infection, Thrombo-embolic complications, Febrile morbidity
Duration of hospital stay | Upto 1 month
  In days

OTHER OUTCOMES:
BMI | Pre operatively
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Abhilasha Agarwal, MS, Principal Investigator — Manipal University

IPD SHARING:
Plan to Share IPD: Undecided
All IPD that underlie results in a publication maybe shared after sponsor approval. Present status - undecided.

REFERENCES:
- [Background] Wu JM, Wechter ME, Geller EJ, Nguyen TV, Visco AG. Hysterectomy rates in the United States, 2003. Obstet Gynecol. 2007 Nov;110(5):1091-5. doi: 10.1097/01.AOG.0000285997.38553.4b. PMID 17978124
- [Background] Garry R, Fountain J, Brown J, Manca A, Mason S, Sculpher M, Napp V, Bridgman S, Gray J, Lilford R. EVALUATE hysterectomy trial: a multicentre randomised trial comparing abdominal, vaginal and laparoscopic methods of hysterectomy. Health Technol Assess. 2004 Jun;8(26):1-154. doi: 10.3310/hta8260. PMID 15215018
- [Background] Hoffman MS, Lynch CM. Minilaparotomy hysterectomy. Am J Obstet Gynecol. 1998 Aug;179(2):316-20. doi: 10.1016/s0002-9378(98)70358-8. PMID 9731832
- [Background] Fanfani F, Fagotti A, Longo R, Marana E, Mancuso S, Scambia G. Minilaparotomy in the management of benign gynecologic disease. Eur J Obstet Gynecol Reprod Biol. 2005 Apr 1;119(2):232-6. doi: 10.1016/j.ejogrb.2004.07.040. PMID 15808386
- [Background] Pelosi MA 2nd, Pelosi MA 3rd. Pelosi minilaparotomy hysterectomy: a non-endoscopic minimally invasive alternative to laparoscopy and laparotomy. Surg Technol Int. 2004;13:157-67. PMID 15744686
- [Derived] Agarwal A, Shetty J, Pandey D, Jain G. Feasibility and Compatibility of Minilaparotomy Hysterectomy in a Low-Resource Setting. Obstet Gynecol Int. 2018 Aug 1;2018:8354272. doi: 10.1155/2018/8354272. eCollection 2018. PMID 30154857